CLINICAL TRIAL: NCT02320383
Title: A Prospective, Multicenter, Phase-II Trial Evaluating Efficacy and Safety of Bendamustine + GA101 (BG) in Patients With Relapsed CLL Followed by Maintenance Therapy With GA101 for Responding Patients
Brief Title: CLLR3: Bendamustine + GA101 (BG) in Relapsed or Refractory CLL Followed by GA101 Maintenance for Responding Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Munich Municipal Hospital (Other)
Collaborators: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLLR3
Record Dates: First submitted 2014-09-01; First posted 2014-12-19 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Chronic Lymphocytic Leucemia
Keywords: CLL
MeSH Terms: interventions — obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- B + GA101 (Experimental): Induction:
  Bendamustine + GA101; a maximum of 6 cycles of BG will be administered; each cycle with a duration of 28 days
  Maintenance:
  GA101 i.v. 1000 mg (flat dose): every 84 days starting on final restaging continued until progression or to a maximum of 2 years
  Interventions: Biological: GA101 (Obinutuzumab); Drug: Bendamustine

INTERVENTIONS:
Biological: GA101 (Obinutuzumab) — Induction
  Cycle 1: d1 - 100 mg, (d1 or) d2 - 900 mg, d8+15 - 1000 mg i.v., q28d
  Cycle 2 - 6: d1 - 1000 mg i.v., q28d
  Maintenance
  GA101 iv 1000 mg (flat dose): every 84 days
  Other Names: Gazyvaro
Drug: Bendamustine — Induction
  Cycle 1: d3+4 (or d2+3) - 70 mg/m² i.v., q28d
  Cycle 2 - 6: d2+3 - 70 mg/m i.v., q28d
  Other Names: Ribomustin; Levact

SUMMARY:
A Prospective, Multicenter, Randomized Phase-Ii Trial Comparing Efficacy And Safety Of Fludarabine + Cyclophosphamide + Ga101 (Fcg) And Bendamustine + Ga101 (Bg) In Patients With Relapsed Or Refractory Cll Followed By Maintenance Therapy With Ga101 For Responding Patients

DETAILED DESCRIPTION:
The type II anti-CD20 antibody GA101 has demonstrated a high efficacy as single agent (ORR 62%) and was well tolerated in previously treated patients with CLL.

Additionally, there is evidence that immunochemotherapy consisting of fludarabine, cyclophosphamide and rituximab (FCR) is active in patients with refractory and relapsed CLL.

Besides FCR, the combination of bendamustine with rituximab (BR) has shown to be active in both relapsed and previously untreated patients with CLL.

In preclinical studies GA101, a glycoengineered, humanized type II anti-CD20 antibody, has shown superior activity compared with type I antibodies.

Therefore, a combination therapy with FC + GA101 (FCG) or B + GA101 (BG) might further improve the therapeutic outcome in relapsed or refractory CLL. The CLLR3 trial was designed to investigate and to compare the efficacy and safety of induction with both immunochemotherapies followed additionally by a maintenance therapy with GA101 for responding patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL in need of treatment according to the iwCLL guidelines
2. Relapsed or refractory disease after at least one, but no more than 3 prior regimens for CLL
3. Medically fit patients without relevant comorbidity, defined as total CIRS score ≤6 (single score < 4 for one organ category)
4. ECOG performance status of 0 - 2
5. Hematology values within the following limits unless cytopenia is caused by the underlying disease, i.e. no evidence of additional bone marrow dysfunction (e.g. myelodysplastic syndrome (MDS), hypoplastic bone marrow due to toxicity of prior therapy):

   1. Absolute neutrophil count ≥1.5 x 109/L
   2. Platelets ≥50 x 109/L and more than 7 days since last transfusion
6. Creatinine clearance >60 ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured after 24 h urine collection
7. Adequate liver function as indicated by a total bilirubin, AST, and ALT ≤2 the institutional ULN value, unless directly attributable to the patient's CLL
8. Negative serological Hepatitis B test (i.e. HBsAg negative and anti-HBc negative, patients positive for anti-HBc may be included if PCR for HBV DNA is negative); negative testing of Hepatitis C RNA; negative HIV test within 6 weeks prior to registration
9. 18 years of age or older
10. Life expectancy >6 months
11. Able and willing to provide written informed consent and to comply with the study protocol procedures

Exclusion Criteria:

1. Detected del(17p) or TP53 mutation
2. Refractoriness to FCR / BR
3. Transformation of CLL to aggressive NHL (Richter's transformation)
4. Known central nervous system (CNS) involvement
5. Evidence of significant uncontrolled concomitant disease
6. Major surgery < 30 days before screening
7. Decompensated hemolytic anemia 28 days before screening
8. Hemolytic cystitis 28 days before screening
9. Patients with a history of confirmed PML
10. Prior treatment with GA101
11. History of prior malignancy, except for conditions as listed below (a-d) and if patients have recovered from the acute side effects incurred as a result of previous therapy:

    1. Malignancies treated with curative intent and with no known active disease present for ≥ 2 years before registration
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease at screening
    3. Adequately treated cervical carcinoma in situ without evidence of disease at screening
    4. Surgically adequately treated low grade, early stage localized prostate cancer without evidence of disease at screening
12. Use of investigational agents or concurrent anticancer treatment within the last 4 weeks before registration
13. Patients with active infection requiring systemic treatment
14. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies and/ or known hypersensitivity to any constituent of the product
15. Hypersensitivity to fludarabine, cyclophosphamide, bendamustine, GA101 and/ or to any of the excipients for example mannitol
16. An individual organ/ system impairment score of 4 as assessed by the CIRS definition limiting the ability to receive an intensive therapy for CLL
17. Legal incapacity
18. Women who are pregnant or lactating
19. Fertile men or women of childbearing potential unless:

    1. surgically sterile or ≥2 years after the onset of menopause
    2. willing to use a highly effective contraceptive method (Pearl Index <1) such as those listed at section 4.2.2 Exclusion criteria during study treatment and for 12 months after end of study treatment
20. Vaccination with a live vaccine within a minimum of 28 days before screening
21. Participation in any other clinical trial which would interfere with the study drug
22. Prisoners or subjects who are institutionalized by regulatory or court order
23. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of two regimens of immunochemotherapy, i.e. Response rates of Fludarabine, Cyclophosphamide plus GA101 (FCG) and Bendamustine plus GA101 (BG), in patients with relapsed or refractory CLL. | The response to the induction phase will be performed 84 days after first dose of last cycle of induction administered
  Efficacy of FCG and/ or BG is confirmed if the ORR is at least 80% (response rate of an active regimen) respectively and is assessed to be not effective if the ORR is 60% or less (ORR of an uninteresting regimen).

SECONDARY OUTCOMES:
MRD levels | MRD levels will be assessed at 84 days after first dose of last cycle of induction and during maintenance every 3 months up to 2 years for responding patients
  MRD levels (evaluation of minimal residual disease (MRD)) by flow cytometry during treatment and maintenance
Progression free survival (PFS) | The time to disease progression will be measured from the date of randomization to the date of first disease progression, assessed up to 54 months
  From the date of randomization to the date of first disease progression (as defined by the iwCLL response criteria) or death by any cause, whichever occurs first.
Event-free survival (EFS) | From the date of randomization to the date of first disease progression, start of next CLL treatment or death by any cause, whichever occurs first, assessed up to 54 months
Overall survival (OS) | Overall survival (OS) will be calculated from the date of randomization to the date of death due to any cause, assessed up to 54 months
Duration of response in patients with CR/ CRi, clinical CR / clinical CRi or nPR/ PR | This will be measured from the date of first documentation of response to the date of first disease progression, or death by any cause, whichever occurs first, assessed up to 54 months
Time to next anti-leukemia treatment | From time of randomization to the date of initiation of next treatment for CLL or death by any cause, whichever occurs first, assessed up to 54 months
Overall response rate in biological defined risk groups | The response to the induction phase will be performed 84 days after first dose of last cycle of induction administered
  Is defined by the proportion of patients having achieved a CR/ CRi, clinical CR/ CRi or nPR/ PR as best response based on the respective population.
Complete response rate | The response to the induction phase will be performed 84 days after first dose of last cycle of induction administered
  Is defined by the proportion of patients having achieved a CR/ CRi as best response based on the respective population (= number of patients with best response CR/ CRi divided by the number of the respective population).
Safety parameters during induction and maintenance phase | SAE: until end of study, AE: From day 1 of the first cycle until 28 days after the end of the treatment, assessed up to 54 months
  During induction and maintenance phase until End of Study. Safety parameters: type, frequency, and severity of adverse events (AEs) and relationship of AEs to study treatment. Furthermore the safety profile including second malignancies of patients treated with FCG/ BG induction treatment and patients with and without maintenance will be evaluated and compared descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens-Martin Wendtner, Prof. Dr., Principal Investigator — Klinikum München GmbH
Locations (1):
- German CLL Study Group, Cologne, Germany